CLINICAL TRIAL: NCT03930823
Title: Advance Care Planning Among Older People From Turkish Origin in Belgium: An Exploratory Interview Study
Brief Title: Interviews With Older People From Turkish Origin in Belgium About Advance Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACP-TR-1-2018
Record Dates: First submitted 2019-04-17; First posted 2019-04-29 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-05

CONDITIONS: Advance Care Planning; Ethnic Minorities; Turkish Origin; Advance Medical Directives; Muslims; Living Will
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: One to one Interviews
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Other): One to one interviews with older people from Turkish origin in Belgium
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — One to one interview

SUMMARY:
Advance care planning (ACP) enables individuals to define goals and preferences for future medical treatment and care, to discuss these goals and preferences with family and health-care providers, and to record and review these preferences if appropriate. Research has shown that most Western patients express the need about what ACP entails.

Ethnicity creates an important cultural impact on how people look at life and death, so that there is an influence on making decisions about end-of-life care. The Turkish ethnic group is one of the largest visible non-Western minority groups in Western countries. Studies on how ACP is perceived among patients from Turkish origin are lacking.

The objective of this study is exploring the knowledge, experiences, point of views, preferences, attitudes, facilitators and barriers concerning advance care planning of older people from Turkish origin in Belgium. Semi-structured interviews (in the native Turkish language) will be used.

ELIGIBILITY:
Inclusion Criteria:

People:

* with Turkish origin who live in Belgium and are older than 65 years
* who have also given informed consent to participate in this qualitative interview study

Exclusion Criteria:

* Patients who are terminal ill which means having a life-limiting disease with irreversible decline and who are actively dying (actively dying is related to patients with days of survival). (41)
* Having cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Knowledge about advance care planning from older people from Turkish origin in Belgium | 9 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: What do you know in relation to advance care planning?
Experiences about advance care planning from older people from Turkish origin in Belgium | 9 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions:Have you yourself ever thought about your future healthcare? Have you yourself ever looked up something about that?
Views/preferences about advance care planning from older people from Turkish origin in Belgium | 9 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: What do you think about discussing advance care planning now for the future? Even if you do not have such a serious illness at the moment, what are the advantages and disadvantages about discussing your wishes for the future, now?
Attitudes about advance care planning from older people from Turkish origin in Belgium | 9 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: Before you got severe illness, do you wish to discuss to someone your future wishes in advance? Why? Do you wish to give authority on your behalf to someone? Why?
Barriers and facilitators for advance care planning from older people from Turkish origin in Belgium | 9 months
  This is a qualitative study. We developed a semi-structured interview guide with the following questions: In your opinion, what makes it easier or what would make it easier to talk about advance care planning? In your opinion, what makes it harder to talk about advance care planning?

CONTACTS AND LOCATIONS:
Overall Officials: Hakki Demirkapu, MD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Faculteit Geneeskunde en Farmacie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No